CLINICAL TRIAL: NCT05588739
Title: Evaluating the Feasibility of a Cognitive-Behavioral Therapy for Children With Nightmares as a Mediator of Suicide Risk
Brief Title: Cognitive-Behavioral Therapy for Children With Nightmares as a Mediator of Suicide Risk (COMAA)
Acronym: COMAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: University of Tulsa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB12343
Record Dates: First submitted 2022-10-03; First posted 2022-10-20 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Nightmare
Keywords: Nightmares; Children; Trauma; CBT; Exposure; Relaxation; Rescripting; Cognitive; Behavioral; Therapy; Suicidality
MeSH Terms: conditions — Wounds and Injuries; Behavior; Suicidal Ideation | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Blinded randomization into 2 groups: Treatment & Waitlist Control. Treatment group receives treatment right away. Waitlist group receives treatment after a 5 week wait.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Right-Away (Experimental): Cognitive Behavioral Therapy using exposure, relaxation, and rescripting - Child utilizes behavioral and cognitive therapy techniques of exposure therapy and cognitive restructuring.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Waitlist Control (No Intervention): Waitlist control group will complete pre and post assessments at beginning and end of wait period.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — The manualized CBT protocol is five session that teach sleep hygiene, relaxation strategies, and addresses nightmares therapeutically through exposure and rescripting.
  Arms: Treatment Right-Away

SUMMARY:
Youth suicide risk has increased 56% in the last decade, and suicide is the leading cause of preventable death in children and adolescents. Experiencing chronic nightmares doubles the risk of suicidal ideation in children and adolescents. Decades of research support that even when controlling for depression and insomnia, nightmares predict suicidality. Contemporary theories model nightmares as the mediating link between depression and suicide. Numerous studies examine the effect of nightmare-specific therapies on reducing suicide in adults, but none have examined whether nightmare therapies can reduce youth suicidality. The proposed pilot will evaluate the feasibility of the Cognitive Behavioral Therapy for Nightmares in Children paradigm (CBT-NC), recruiting and retaining children ages 6-17 who experience chronic nightmares. Utilizing a waitlist control (WL) model, participants (n=30) will be randomized after baseline assessment to either immediate treatment or a WL. Feasibility will be evaluated by examining retention through treatment (or WL) to post WL and post treatment assessments. Both groups will be evaluated before and after the treatment for suicidal ideation, sleep quality, and nightmare distress and frequency, in order to document improvements due to therapy. The proposed pilot will provide preliminary data about recruitment, retention, and allow for effect size calculations between groups. These results will be used to develop a larger treatment study that would ultimately evaluate the mediating effect of treatment for chronic nightmares on suicidality in children.

ELIGIBILITY:
Inclusion Criteria:

* Child must be between the ages of 6-17 years 11 months.
* Child must report recurrent nightmares that meet DSM criteria for nightmare disorder.
* Child must speak and understand English at no less than a 6 year old level.
* Children on prescribed psychotropic medications must be stable for 30 days prior to enrolling.
* Child must have a parent or legal guardian attend study visits with them.
* Participants must have access to WIFI/phone data in order to participate in this study, and must have an electronic device with a camera enabled. Our study team will have the capability of driving a tablet to the participant's home if that is the only reason they cannot participate, and if the family lives within the greater Tulsa area.

Exclusion Criteria:

* Children with a previous diagnosis of sleep apnea which is not adequately treated.
* Children whose receptive/expressive language skills are below a 6 year old level.
* If it is determined that a child is actively suicidal and at imminent risk for self-harm, the family will be notified and referred for immediate care. They will not be eligible for the study until they are deemed stable.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Change on the Child Adolescent Trauma Screen (CATS) - Child Version | Participants will be assessed at Baseline (Week 0) through study completion, up to 15 weeks.
  The CATS screens for child trauma history and PTSD symptoms in youth ages 7-17; 15 YES/NO questions; 1 open-ended question
Change on the Trauma Related Nightmare Survey - Child Version (TRNS-C) | Participants will be assessed at Baseline (Week 0) through study completion, up to 15 weeks.
  The TRNS-C is a 14 item self report questionnaire that assesses current sleep quality, frequency, severity, and duration of nightmares, as well as cognitions, emotions, and behaviors related to nightmares in children.
Change on Sleep Locus of Control (SLOC) | Participants will be assessed at Baseline (Week 0) through study completion, up to 15 weeks.
  The SLOC is an 6 item self report measure perceived contingencies between sleep behavior and events. This scale is collected as a child self report, and a caregiver report regarding child.
Change on Nightmare Locus of Control (NLOC) | Participants will be assessed at Baseline (Week 0) through study completion, up to 15 weeks.
  The N-LOC is an 6 item self report. This scale is collected as a child self report, and a caregiver report regarding child.
Change in reports on Sleep Journal | Participants complete this assessment at Pre-treatment (for 1 week), daily during the treatment phase (an average of 5 weeks), at Post treatment (for 1 week).
  6 question self report that patient assesses daily from home.
Change on the Child Adolescent Trauma Screen (CATS) - Caregiver Report regarding child | Participants will be assessed at Baseline (Week 0) through study completion, up to 15 weeks.
  The CATS screens for child trauma history and PTSD symptoms (information obtained from the caregiver, about the child).
Change on Center for Epidemiologic Studies Beliefs and Attitudes About Sleep Scale (DBAS-16) | Participants will be assessed at Baseline (Week 0) through study completion, up to 15 weeks.
  The DBAS-16 is a 16-item self-report measure that evaluates the role of sleep related beliefs. The score is a sum of the 16 items, ranging from 16 to 80. Higher scores represent more dysfunctional beliefs about sleep.
Change on Center for Epidemiologic Studies Depression Scale for Children (CES-DC) | Participants will be assessed at Baseline (Week 0) and after post-condition (Week 6).
  The CES-DC is a 20-item self-report depression inventory. A score of 15 or higher indicates significant levels of depression.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Tulsa, Tulsa, Oklahoma
  - University of Oklahoma School of Community Medicine, Tulsa, Oklahoma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cromer LD, Bell SB, Prince LE, Hollman N, El Sabbagh E, Buck TR. Efficacy of a telehealth cognitive behavioral therapy for improving sleep and nightmares in children aged 6-17. Front Sleep. 2024 Jul 11;3:1401023. doi: 10.3389/frsle.2024.1401023. eCollection 2024. PMID 41424486